CLINICAL TRIAL: NCT05443685
Title: An Open-Label, Phase 1/2, Single-Site Study of the Safety, Biochemical Efficacy, and Exploratory Clinical Effects of Oral ADX-629 in Subjects With Sjögren-Larsson Syndrome
Brief Title: ADX-629 Therapy for Sjogren-Larsson Syndrome
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0517-22-FB; SLS-ADX-629-001 (Other: commercial sponsor)
Record Dates: First submitted 2022-06-10; First posted 2022-07-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-03

CONDITIONS: Sjogren-Larsson Syndrome
Keywords: ichthyosis; spasticity; intellectual disability; retinopathy; spastic diplegia
MeSH Terms: conditions — Sjogren-Larsson Syndrome; Ichthyosis; Muscle Spasticity; Intellectual Disability; Retinal Diseases; Cerebral Palsy | interventions — ADX-629

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADX-629 treatment (Experimental): Open label treatment with ADX-629
  Interventions: Drug: ADX-629

INTERVENTIONS:
Drug: ADX-629 — Particpants 10-50 years old will be administered ADX-629 250 mg tablets twice daily.
  Participants 5-9 years old will be administered ADX-629 125 mg tablets twice daily.
  Other Names: Open label

SUMMARY:
This research study will determine whether orally administered ADX-629 is safe and has biochemical efficacy in participants with Sjögren-Larsson syndrome (SLS), a rare inherited disorder of fatty aldehyde metabolism The disease is caused by bi-allelic mutations in ALDH3A2, which results in deficient activity of fatty aldehyde dehydrogenase (FALDH) and leads to the build-up of harmful long-chain (C16-C20) aldehydes and alcohols. Accumulation of these lipids and their metabolic products in skin, brain and eyes is responsible for the symptoms, which persist lifelong. ADX-629 is an aldehyde trapping agent that is expected to eliminate fatty aldehydes and negate aldehyde toxicity, improve the biochemical abnormalities and have clinical efficacy for SLS.

The primary objective of this clinical protocol is to determine whether ADX-629 is safe and tolerable for use in SLS subjects. The secondary objective is to determine the efficacy of ADX-629 in reversing the biochemical abnormalities in SLS. Exploratory objectives are to evaluate the short-term clinical effects of ADX-629 on neurologic, cutaneous and ophthalmologic disease in SLS. Participants will be treated with ADX-629 for 12 weeks and monitored for safety and biochemical efficacy.

DETAILED DESCRIPTION:
Sjögren-Larsson syndrome (SLS) is a rare inherited disorder of fatty aldehyde metabolism characterized by congenital ichthyosis, spastic diplegia, intellectual disability, seizures and a distinctive retinopathy. The disease is caused by bi-allelic mutations in ALDH3A2, which results in deficient activity of fatty aldehyde dehydrogenase (FALDH) and leads to the build-up of harmful long-chain (C16-C20) aldehydes and alcohols. Accumulation of these lipids and their metabolic products in skin, brain and eyes is responsible for the symptoms, which persist lifelong. Investigators hypothesize that elimination of fatty aldehydes using the oral pharmacologic aldehyde trapping agent ADX-629 will negate aldehyde toxicity, improve the biochemical abnormalities and have clinical efficacy for SLS patients.

This study is an open label, Phase 1/2, single center investigation of ADX-629 in SLS. The primary objective is to determine whether ADX-629 is safe and tolerable for use in SLS participants. The secondary objective is to determine the efficacy of ADX-629 in reversing the biochemical abnormalities in SLS. Exploratory objectives are to evaluate the short-term clinical effects of ADX-629 on neurologic, cutaneous and ophthalmologic disease in SLS.

Up to 10 paticipants with genetically confirmed SLS who meet eligibility criteria will be enrolled. All participantss will be studied at the University of Nebraska Medical Center/Children's Hospital & Medical Center in Omaha, Nebraska. Participants will be treated with ADX-629 administered orally as 250 mg tablets for 12 weeks. Participants will be monitored for safety of ADX-629 every 4 weeks by physical examination and biochemical safety tests.

The effects of ADX-629 on SLS-specific biomarkers will be determined after 12 weeks of drug treatment. Clinical tests will monitor neurological, dermatological and ophthalmologic response to drug.

ELIGIBILITY:
Inclusion Criteria:

* Patricipant or participant's guardian is willing to provide written informed consent prior to the initiation of any study procedures. Assent will be solicited from participant intellectually capable of providing assent.
* Participant is willing to comply with all study procedures and availability for the duration of the study.
* Participant is 5-50 years of age at the time of enrollment.
* Participant has a genetically-confirmed diagnosis of SLS with two pathogenic sequence variants in ALDH3A2.
* Participant has active ichthyosis and neurologic symptoms of spasticity.
* Participant is able to swallow oral tablet medication and is willing to adhere to the study regimen.
* Participant is willing to suspend use of all topical creams 7 days before initial baseline evaluation and before the 12-week center visit.
* Participant has not been treated with any experimental drug for 1 month before baseline visit and during ADX-629 treatment.
* Participant who is sexually active agrees to use adequate contraception throughout the duration of the study, as follows:
* For females of child-bearing potential: Negative pregnancy test at Baseline and compliant with a medically approved contraceptive regimen during the study or documented to be surgically sterile or postmenopausal.
* For sexually-active men: Compliant with a barrier contraceptive regimen during the study.

Exclusion Criteria:

* History of any malignancy within 5 years of screening except for basal cell or squamous cell in situ skin carcinomas or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
* Participant is known to be human immunodeficiency virus (HIV) positive or has other known immunodeficiency.
* Participant has evidence of an active systemic or skin infection, including severe acute respiratory syndrome (SARS-CoV-2).
* History of significant tachycardia, bradycardia, acute or chronic cardiovascular disease, or any clinically significant abnormalities in rhythm or conduction detected on electrocardiogram (ECG), or QT interval corrected for heart rate using Fridericia's formula (QTcF) of >440 ms or <340 ms during screening.
* History or presence of gastrointestinal, hepatic disease, moderate or severe hepatic impairment (defined as Child-Pugh Class B and Class C) or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drug.
* Acute or chronic renal disease, moderate or severe renal impairment, history of renal disease, or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 calculated by Chronic Kidney Disease Epidemiology (CKD-EPI) equation.
* History of any other condition that, in the opinion of the Investigator, would compromise the participant's ability to comply with the protocol or that might compromise the participant's safety or the interpretation of the study results.
* Participant is currently receiving immunosuppressive therapy, including intermittent or low-dose corticosteroids and is not able or willing to suspend its use for a period from 2 weeks before and throughout the study.
* Participant is currently receiving and refuses to interrupt any systemic or topical medication that is excluded.
* Participant received an investigational systemic or topically administered prescription drug within 30 days before enrollment.
* Participant has received botulinum toxin (Botox) injections within 6 months of enrollment.
* Participant has a known allergic reaction to any ingredients of study drug formulation.
* Participant is currently participating in any other therapeutic clinical study.
* Participant is pregnant, intending to become pregnant, or breastfeeding.

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0 | weekly for 12 weeks
  Participants are required to report any adverse events as they arise and will be contacted weekly for information regarding adverse events. Physical examinations with vital signs will be done monthly.
Number of Participants With Abnormal Drug-related Safety Blood Tests | monthly for 12 weeks
  Participants will have monthly medical tests to monitor safety of ADX-629 including complete blood count, comprehensive chemistry panel, vitamin A, vitamin B6 (pyridoxal phosphate), homocysteine, and urinalysis.
Compliance and Tolerability of ADX-629 | daily for 12 weeks
  A written drug log will be required for recording daily administration of ADX-629 tablets and any problems tolerating the drug. Unused tablets will be counted as a measure of compliance.

SECONDARY OUTCOMES:
Biochemical Efficacy of ADX-629 as Determined by Reversal of Abnormal Biomarkers | Tests will be done at week 1 and week 12.
  Biochemical efficacy of ADX-629 in reversing disease-specific abnormalities in blood levels of fatty alcohols, alkylglycerol lipids, SLS metabolomic profile, SLS lipid profile, and oxidative stress markers. Skin elasticity and thickness, transepidermal water loss, stratum corneum fatty alcohols and alkylglycerol lipids will also be measured.

OTHER OUTCOMES:
Exploratory Clinical Outcomes to Determine Drug Dependent Changes in Abnormal Clinical Measures | Examinations and procedures will be done at week 1 and week 12.
  Clinical response to ADX-629 will be determined with brain MRI, magnetic resonance spectroscopy, EEG, clinical spasticity scores, visual index of ichthyosis severity score, and SLS retinopathy based on eye exam and retinal photographs.

CONTACTS AND LOCATIONS:
Overall Officials: William B Rizzo, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate de-identified data will be shared with other investigators by request.

REFERENCES:
- [Background] Rizzo WB. Sjogren-Larsson syndrome: molecular genetics and biochemical pathogenesis of fatty aldehyde dehydrogenase deficiency. Mol Genet Metab. 2007 Jan;90(1):1-9. doi: 10.1016/j.ymgme.2006.08.006. Epub 2006 Sep 22. PMID 16996289
- [Background] Rizzo WB. Genetics and prospective therapeutic targets for Sjogren-Larsson Syndrome. Expert Opin Orphan Drugs. 2016 Apr;4(4):395-406. doi: 10.1517/21678707.2016.1154453. Epub 2016 Mar 10. PMID 27547594
- [Background] Rizzo WB, S'aulis D, Dorwart E, Bailey Z. Sjogren-Larsson syndrome: A biochemical rationale for using aldehyde-reactive therapeutic agents. Mol Genet Metab Rep. 2021 Dec 23;30:100839. doi: 10.1016/j.ymgmr.2021.100839. eCollection 2022 Mar. PMID 35242571